CLINICAL TRIAL: NCT06381609
Title: Contribution of Addiction Peer Support on Adherence to Care and Clinical Outcomes in Alcohol Dependence: a Prospective Controlled Trial With Medico-economic Component
Brief Title: Peer Support in Alcohol Dependence
Acronym: PEERSIAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL22_0901
Record Dates: First submitted 2024-04-02; First posted 2024-04-24 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Use Disorder
Keywords: Peer support; Addiction; Alcohol
MeSH Terms: conditions — Alcoholism; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer support Group (Experimental): 313 patients will be recruited over 3 years in the peer support group. Patients will be accompanied by an addiction peer support specialist, as part of an "add-on" follow-up compared with conventional follow-up (same management as in the control group).
  Interventions: Behavioral: Quality life questionnaire AQoLS; Behavioral: Quality life questionnaire Euroqol EQ-5D-5L; Other: Peer support consultations
- Control Group (Active Comparator): 313 patients will be recruited over 3 years in the control group. Patients will receive "as usual" outpatient abstinence-maintenance follow-up, with consultations of all kinds (medical, psychological, nursing, group, etc.)
  Interventions: Behavioral: Quality life questionnaire AQoLS; Behavioral: Quality life questionnaire Euroqol EQ-5D-5L

INTERVENTIONS:
Behavioral: Quality life questionnaire AQoLS — Quality life questionnaire AQoLS will be completed by patients of both arms at inclusion, three and six months after inclusion
Behavioral: Quality life questionnaire Euroqol EQ-5D-5L — Quality life questionnaire Euroqol EQ-5D-5L will be completed by patients of both arms at inclusion, three and six months after inclusion
Other: Peer support consultations — For patients included in the Peer support group, eight mandatory consultations with a peer support specialist will be performed between the inclusion visit and during the three following months.
  Patients can request additional consultations with the peer support specialist during the 6 first months of follow-up
  Arms: Peer support Group

SUMMARY:
Alcohol use disorder (AUD) affects between 4% and 6% of French adults, and requires appropriate medical treatment.

However, 20-40% of patients with AUD are lost to follow-up at an early stage. Consequently, it is important for addiction departments to implement and evaluate innovative tools and interventions, including the involvement of peer support, to help patients remain in care, and to assess whether peer support has a positive impact on their clinical outcome.

Addiction peer support specialists (APSSs) are individuals who have personally experienced addiction, and who have decided to use their experience to assist other people going through a similar situation, after completing a specific official graduation.

Compared to other caregivers, APSSs may induce in patients a sense of identification which could improve the patient motivation to engage and remain in care.

This is the main hypothesis and the main scientific objective of the PEERSIAD study, which will aim to confirm that accompanying patients with AUD using APSSs after alcohol detoxification, reduces the rate of lost-to-follow-up and improves the overall clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18
* Socially insured
* Meeting DSM-5 criteria for alcohol use disorder (AUD)
* Abstinent from alcohol and involved in supervised alcohol withdrawal for at least 5 days and no more than 21 days (outpatient or inpatient)
* Starting a post-detoxification outpatient program

Exclusion Criteria:

* Other severe substance use disorder, i.e. DSM-5 criteria ≥ 6 (excluding tobacco)
* Patient under protective measure (safeguard measure, guardianship) or deprived of liberty or in ordered care and hospitalization measures without consent.
* Inability to communicate and express oneself orally in French, compromising the possibility of exchanges between the Peer support and the patient.
* Psychiatric or cognitive comorbidities making inclusion impossible, at the investigator's discretion.
* Individual accompaniment by a Peer support in the 15 days prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Unplanned cessation of care at 6 months | At 6 months after inclusion
  The unplanned cessation of care at 6 months, excluding consultations with an APSS, with no further contact in the following month, is defined as having had a last planned consultation that was not fulfilled between M0 and M6

SECONDARY OUTCOMES:
Number of unfulfilled consultations | 6 months after inclusion
  The number of unfulfilled consultations (scheduled consultations, excluding Peer Support consultations, without patient's visit with or without justification) over the 6-month study follow-up period, collected from the medical records of the addictology department.
Euroqol-5D-5L questionnaire score | At inclusion, 3 and 6 months after inclusion
  The differential cost-utility ratio, in relation to the innovative strategy including a Peer Support, will be assessed using the Euroqol-5D-5L questionnaire (EQ-5D-5L).
Difference in costs (in euros) | At 1, 2 and 3 years after the beginning of implementation on French territory
  An additional analysis will be carried out if the cost-utility ratio is positive: Difference in costs (in euros) for the payer (French compulsory health insurance) between a scenario in which the innovative management is implemented and disseminated in practice and on French territory, and a scenario in which usual follow-up is maintained.
Number of AUD criteria according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) | At inclusion, 3 and 6 months after inclusion
Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) score | At inclusion, 3 and 6 months after inclusion
average number of standard drinks declared per week | At inclusion, 3 and 6 months after inclusion
Alcohol Quality of Life Scale (AQoLS) score | At inclusion, 3 and 6 months after inclusion
  Changes in quality of life will be measured using the AQoLS
State-Trait Anxiety Inventory (STAI-Y) score | At inclusion, 3 and 6 months after inclusion
  Changes in levels of anxiety will be measured using STAI-Y
Montgomery-Åsberg Depression Rating Scale (MADRS) score | At inclusion, 3 and 6 months after inclusion
  Changes in levels of depression will be measured using MADRS
Cannabis Use Disorders Identification Test - Revised (CUDIT-R) score | At inclusion, 3 and 6 months after inclusion
  Changes in the severity of cannabis use will be measured by the CUDIT-R score
type of opioid use | At inclusion, 3 and 6 months after inclusion
frequency of opioid use | At inclusion, 3 and 6 months after inclusion
type of psychostimulant use | At inclusion, 3 and 6 months after inclusion
frequency of psychostimulant use | At inclusion, 3 and 6 months after inclusion
Fagerström test score | At inclusion, 3 and 6 months after inclusion
  Tobacco use will be measured by the Fagerström test
Health Care Satisfaction Questionnaire (HCSQ) score | At 6 months after inclusion
  Patient's satisfaction will be measured by HCSQ questionnaire
Number of hospitalisations | At 6 months after inclusion
  Measurement of the number of hospitalisations related or not to the AUD and the ratio of total hospital days to number of hospital admissions (based on medical records and patient interviews)
Service organization description | Before setting up of the study
Description of type of support and missions performed by Peer Support | After last visit of last patient (around 3,5 years after first inclusion)
Acceptability of Intervention Measure (AIM) score | After last visit of last patient (around 3,5 years after first inclusion)
  AIM score measured in Peer Support and medical staff
AIM score | At 6 months after inclusion
  AIM score measured in patients
Adoption of intervention | After last visit of last patient (around 3,5 years after first inclusion)
  adoption of intervention will be assessed through semi-structured interviews and measurement of the number of patients followed-up versus the number of eligible patients, refusals to be accompanied by APSS, and premature discontinuation of follow-up
Intervention fidelity | After last visit of last patient (around 3,5 years after first inclusion)
  intervention fidelity will be assessed by monitoring APSS activity indicators, describing deviations from the protocol and semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin ROLLAND, Principal Investigator — Hopsices Civils de Lyon
Locations (5):
- France (5):
  - CH Le Vinatier, Bron
  - Hôpital Beaujon, Clichy
  - GH Nord, Hospices Civils de Lyon, Lyon
  - CHS St Anne, Paris
  - Bichat Hospital, Paris

IPD SHARING:
Plan to Share IPD: No